CLINICAL TRIAL: NCT03029897
Title: Impact of E-reporting by Patients With Relapsing-remitting Multiple Sclerosis on the Reporting of Adverse Drug Reactions in France: a Randomized Controlled Trial.
Brief Title: E-reporting of Adverse Drug Reactions by Patients in Relapsing-remitting Multiple Sclerosis
Acronym: VigiP-SEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16-135
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Last update posted 2019-07-02 (Actual); Status verified 2018-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: clusters
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): Patients are educated on the use of a mobile application to report adverse drug reactions
  Interventions: Other: My eReport France
- control (No Intervention): Patients are not educated on the use of a mobile application to report adverse drug reactions

INTERVENTIONS:
Other: My eReport France — patients are educated to the use of "My eReport France" application
  Arms: experimental

SUMMARY:
Adverse drug reactions are collected exhaustively during the experimental development phase of the drug, but the trial population is not representative. In post-marketing authorization, the use in the real life of medicines requires to specify the profile of adverse effects through pharmacovigilance. However, in clinical practice, under-reporting of adverse drug reactions prevents a satisfactory knowledge of the risks. For example, in the multiple sclerosis (MS) patients population in 2015, only 1 case of congestive flushing was reported by physicians, none by patients, for approximately 7,800 patients treated with Tecfidera® dimethyl-fumarate, while trials reported 39% of flush.

The investigators propose a study measuring the impact of the deployment of e-reporting to patients in a population suffering from multiple sclerosis in initiation of first line drug therapy. The study design will be a randomized controlled trial. Twenty-four direct or indirect partner centers of the OFSEP will be randomized in 2 arms (1 standard arm without intervention, and one interventional arm), Each arm including 6 CHU, 3 CHG and 3 liberal neurologists. CHUs will include 10 patients in 6 months, and CHGs and liberal neurologists 5 patients, a total of 180 patients will be included. The expected duration of this study is 12 months, 6 months of inclusion of patients, and one 6-month follow-up period for each patient. At 1 month (+/- 15 days) of the follow-up period of each patient, a questionnaire will be made by telephone call to each patient.

The study is part of the pharmacovigilance system in place in France and aims to improve its efficiency by increasing declarations and therefore earlier detection of signals in order to prevent and minimize risks.

The comparison of the two arms should make it possible to decide on the usefulness of national support for e-reporting, while respecting a good integration with the French pharmacovigilance system.

ELIGIBILITY:
Inclusion Criteria:

Patient (> 18 years) with relapsing-remitting multiple sclerosis. Initiation of treatment of 1st line: interferon β, peginterferon β, glatiramer acetate, teriflunomide, dimethyl-fumarate.

Exclusion Criteria:

Patient with progressively progressive secondary or multiple sclerosis. Patient suffering from multiple sclerosis not treated with a first line treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
number of reports of adverse drug reactions | 6 months
  number of reports of adverse drug reactions per patient in the intervention arm using mobile versus standard arm.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Defer G, Fedrizzi S, Chevanne D, Montastruc F, Briant AR, Parienti JJ, Peyro-Saint-Paul L; French VigipSEP Study Group; Societe Francophone de la Sclerose en Plaques (SFSEP). Adverse Drug Reaction Reporting Using a Mobile Device Application by Persons with Multiple Sclerosis: A Cluster Randomized Controlled Trial. Drug Saf. 2021 Feb;44(2):223-233. doi: 10.1007/s40264-020-01009-z. Epub 2020 Oct 13. PMID 33048319
- [Derived] Defer G, Le Caignec F, Fedrizzi S, Montastruc F, Chevanne D, Parienti JJ, Peyro-Saint-Paul L. Dedicated mobile application for drug adverse reaction reporting by patients with relapsing remitting multiple sclerosis (Vigip-SEP study): study protocol for a randomized controlled trial. Trials. 2018 Mar 9;19(1):174. doi: 10.1186/s13063-018-2560-4. PMID 29523169